CLINICAL TRIAL: NCT05545020
Title: Trivalent Chromium as a Treatment for Rheumatoid Arthritis Patients
Brief Title: Trivalent Chromium Treatment for Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sally Saad Saad Hassouna, Lecturer of Internal Medicine department, Rheumatology and Immunology Unit, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trivalent chromium treatment; 040457 (Registry Identifier: Ethics committee of Faculty of Medicine, Alexandria university, Egypt)
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trivalent chromium (Active Comparator): A dietary supplement already available in market one of its known uses is to control diabetes.
  Interventions: Drug: Trivalent chromium versus synthetic and/ or biological DMARDs
- Immunesuppressants (Active Comparator): Synthetic and/ or biological DMARDs
  Interventions: Drug: Trivalent chromium versus synthetic and/ or biological DMARDs

INTERVENTIONS:
Drug: Trivalent chromium versus synthetic and/ or biological DMARDs — Supplement and immunesuppressants
  Other Names: Pure trivalent chromium (not in the form of a compound) and treatments the patients are already taking in comparison

SUMMARY:
Trivalent chromium has shown good results in abolishing inflammation and had a successful result in treating animal model of rheumatoid arthritis. In addition to that, trivalent chromium lacks many side effects which are related to the already known medications of the disease.

So this study aims to evaluate the efficacy of trivalent chromium supplementation in rheumatoid arthritis treatment and measuring the outcomes of that in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a debilitating autoimmune disease which is treated by medications that have many side effects. Trivalent chromium, a naturally occurring element with regulatory effects on blood sugar, has shown anti-inflammatory properties in many studies and has shown a good response at alleviation of rheumatoid arthritis in the disease animal model. For these reasons trivalent chromium should be tried in rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis

Exclusion Criteria:

* other autoimmune diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Arthritis scored by DAS28 score | three months
  DAS 28 is a score of arthritis
ESR in mm/hr | three months
  lab measures for disease activity
CRP mg/dL | three months
  lab measures for disease activity
Radiological investigations if required (X-RAY, ultrasound, MRI, bone scan) | three months
  To assess joints and bone

SECONDARY OUTCOMES:
Serum urea | three months
  A renal function test to exclude trivalent chromium side effects.
serum creatinine | three months
  A renal function test to exclude trivalent chromium side effects.
SGOT | three months
  A liver function test to exclude trivalent chromium side effects.
SGPT | three months
  A liver function test to exclude trivalent chromium side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria University, Egypt, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassouna SS, Sheta E, Zaki I, Harby SA, Allam EA. Trivalent chromium supplementation ameliorates adjuvant induced rheumatoid arthritis through up-regulation of FOXP3 and decrease in synovial Cathepsin G expression. Inflammopharmacology. 2022 Dec;30(6):2181-2195. doi: 10.1007/s10787-022-01025-8. Epub 2022 Jul 13. PMID 35829940
- [Derived] Hassouna SS, Abdel-Moniem OM. Trivalent chromium versus baricitinib for rheumatoid arthritis treatment: first phase 2/3 randomized controlled trial, is trivalent chromium the upcoming immune-modulator? Inflammopharmacology. 2024 Oct;32(5):3163-3179. doi: 10.1007/s10787-024-01515-x. Epub 2024 Jul 19. PMID 39030450